CLINICAL TRIAL: NCT05769218
Title: PrEP and MOUD Rapid Access for Persons Who Inject Drugs: The CHORUS+ Study
Acronym: CHORUS+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Victory Programs Mobile Prevention Services Van and Navigation Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-43487; R01DA058367 (NIH)
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use Disorder
Keywords: Medication for opioid use disorder; Human immunodeficiency (HIV); Pre-exposure prophylaxis (PrEP); Peer recovery coaching (PRC); Motivational interviewing (MI); HIV self testing; People who inject opioids (PWIO)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — chorus protein, Arabidopsis; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHORUS+ (Experimental): The baseline questionnaire for participants in this arm will be followed by a 30-minute motivational interviewing (MI) session with the peer recovery coach (PRC), and will assess readiness for change and provide information about PrEP. The PRC will also assess readiness for MOUD, and this will be further explored during subsequent visits.
  Interventions: Behavioral: CHORUS+
- Usual care- control (Active Comparator): Participants in this arm will receive passive referral for care. there will be no PRC MI session and they will not be offered PrEP or MOUD.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: CHORUS+ — The CHORUS+ intervention will include a baseline interview with a peer recovery coach to encourage uptake of HIV PrEP (pre-exposure prophylaxis) and medications for opioid use disorder (MOUD) through motivational interviewing (MI). Participants will also be offered HIV self-testing on the day of recruitment, HIV PrEP (if they are HIV negative) and MOUD. Participants will then receive peer coaching for 6 months to increase adherence to PrEP and or MOUD.
  Arms: CHORUS+
Other: Standard of care — Normal protocols for care of participants who inject opioids will be followed.
  Arms: Usual care- control

SUMMARY:
The US opioid overdose epidemic has been accompanied by an increase in human immunodeficiency (HIV) among persons who inject drugs. HIV pre-exposure prophylaxis (PrEP) is an FDA approved medication taken daily orally by individuals who are HIV negative, but who are at increased risk for HIV. In order to obtain PrEP, a prescription is needed. Before being prescribed HIV PrEP, it is recommended by the Centers for Disease Control and Prevention (CDC) to obtain an HIV test first. Although home HIV self-test kits are recommended by the CDC and are locally available, uptake remains low.

CHORUS+ (Comprehensive HIV, Hepatitis C, and Opioid Use Disorder Response to the Unaddressed Syndemic +) is a theory-based, peer-delivered, mobile phone-supported intervention focused on enhancing uptake and adherence to HIV PrEP (primary outcome), and continuation of MOUD (secondary outcome) among persons who inject opioids. At recruitment, the intervention will include HIV self-testing, rapid initiation of PrEP and MOUD, and 6-month peer recovery coaching (PRC) to support adherence to these medications. This research study seeks to determine the efficacy of a novel intervention to increase the uptake of evidence-based measures to prevent HIV and treat opioid use disorder.

The efficacy of this multi-site, two-arm randomized control trial of CHORUS+ and usual care [passive referral]. This study is not testing the efficacy of PrEP or HIV home testing which is already known. In addition the investigators will determine the influence of HIV self-testing on PrEP uptake and adherence. In the CHORUS+/ intervention arm, there will be a baseline in-person session with the participant to encourage uptake of PrEP and MOUD using motivational interviewing (MI).

ELIGIBILITY:
Inclusion Criteria:

* Injected opioids within the past 6 months (by self-report)
* Willingness to provide contact information for two family members or friends
* Willingness to sign medical records release forms
* Ability to speak English
* Plans to reside in Boston area for the next 6 months

Exclusion Criteria:

* Individuals with HIV (self report)
* Express desire to harm themselves or others
* Individuals who are pregnant at baseline
* Individuals who are already enrolled in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to HIV PrEP at 6 months Adherence to HIV PrEP | 6 months
  This outcome will be assessed by the proportion of individuals who have dried blood spot tenofovir-diphosphate (TFV-DP) blood level 700 fmol/punch or greater at 6 months post-enrollment.

SECONDARY OUTCOMES:
Adherence to PrEP at 3 and 12 months | 3 months. 12 months
  Adherence will be assessed by self-report and chart review of active medication refills for PrEP and appointments attended.
Receipt of medication for opioid use disorder (MOUD) | 3 months, 6 months, and 12 months
  Receipts will be assessed by any of the following: (1) chart review of active medication refills for MOUD, (2) self-report, (3) urine toxicology results checked during study visit, and (4) chart review for appointments attended.
Test results for gonorrhea | Baseline, 3 months, 6 months, and 12 months
  Results will be assessed as negative or positive.
Test results for chlamydia | Baseline, 3 months, 6 months, and 12 months
  Results will be assessed as negative or positive.
Test results for syphilis | Baseline, 3 months, 6 months, and 12 months
  Results will be assessed as negative or positive.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina A Assoumou, MD MPH, Principal Investigator — Boston Medical Center, Infectious Diseases
Locations (2):
- United States (2):
  - Boston Medical Center Faster Paths Bridge Clinic, Boston, Massachusetts
  - Victory Programs Mobile Prevention Services Van and Navigation Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller SE, Dukes KA, Damato-MacPherson C, Psaros C, Scott NA, Taylor JL, Muroff J, Winter MR, Skiba LE, Lugo H, Cruz R, Ruiz-Mercado G, Crawford ND, Mayer KH, Assoumou SA. Pre-exposure prophylaxis (PrEP) and medications for opioid use disorder for persons who inject drugs: the CHORUS + randomized controlled trial study protocol. Addict Sci Clin Pract. 2025 Dec 25;21(1):17. doi: 10.1186/s13722-025-00634-2. PMID 41449454